CLINICAL TRIAL: NCT05743205
Title: A Pilot Intervention Study to Promote Wellness in Advanced Practice Providers (APPs)
Brief Title: Advanced Practice Provider Intervention Study to Promote Wellness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colleen J Klein (Other)
Responsible Party: Sponsor-Investigator, Colleen J Klein, Education and Research Scientist, OSF Healthcare System
Organization: OSF Healthcare System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1537818
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Job Stress; Professional Burnout
Keywords: Resilience; Burnout; Work engagement
MeSH Terms: conditions — Occupational Stress; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention (Experimental): Educational intervention
  Interventions: Behavioral: voluntary consultative wellness session

INTERVENTIONS:
Behavioral: voluntary consultative wellness session — Professional wellness counseling sessions provided to health care professionals through voluntary enrollment. Consultative sessions will conducted throughout the course of 1 year and number of subsequent sessions will be determined by the participant.

SUMMARY:
This exploratory pilot study is designed as interventional study to examine the efficacy of a wellness initiative that involves use of a licensed clinical professional counselor (LCPC) to assist in the development of diverse coping strategies such as management of stressors, self-care, time management, and any other goals, problems or concerns that APPs would like assistance with during the intervention period.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate an educational professional wellness program designed to assist professional clinicians in developing self-awareness and self-care choices as a means to improve engagement and resilience and to avoid/reduce burnout.

ELIGIBILITY:
Inclusion Criteria:

* employment within non-profit health care setting as a health care professional
* working at least 50% of time in direct patient care
* availability and interest in initial and follow-up wellness visits

Exclusion Criteria:

* actively participating in formalized counseling sessions through other services at time of recruitment into the study

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Holmes-Rahe Life Stress Inventory; The Social Readjustment Rating Scale | change from baseline stress measure at 1 year and 2 years.
  The Holmes-Rahe Scale is used to life changes that may impact stress. Minimum values =150 pts or less; maximum values = 300 pts. or more; higher scores indicate higher susceptibility to stress-induced health problems.
The Brief Resilience Scale | change from baseline in resilience measure at 6 months, 1 year and 2 years.
  The Brief Resilience Scale developed by Smith et al. (2008) is used to measure resilience. Minimum value =6 and maximum value = 30; mean value is used to determine scoring with higher value indicating more resilience.
The Work and Well-being Survey (UWES)© Engagement Scale | change from baseline engagement measure at 6 months, 1 year and 2 years.
  Work engagement is measured using the Utrecht Work and Well-being Survey Engagement instrument (UWES). The minimum value =0 and the maximum value = 54. Mean is used to determine scoring. Higher value indicates greater work engagement.
Advanced Practice Provider Well-being Index | change from baseline well-being measure at 6 months, 1 year and 2 years.
  measures the increased probability of distress risk for personal or professional consequences. Minimum value =0 and maximum value =7. Mean and standard deviation is computed and compared to normative data.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Klein, PhD, RN, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF HealthCare System, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein CJ, Weinzimmer LG, Cooling M, Lizer S, Pierce L, Dalstrom M. Exploring burnout and job stressors among advanced practice providers. Nurs Outlook. 2020 Mar-Apr;68(2):145-154. doi: 10.1016/j.outlook.2019.09.005. Epub 2019 Nov 8. PMID 31708107
- [Background] Klein CJ, Dalstrom M, Lizer S, Cooling M, Pierce L, Weinzimmer LG. Advanced Practice Provider Perspectives on Organizational Strategies for Work Stress Reduction. West J Nurs Res. 2020 Sep;42(9):708-717. doi: 10.1177/0193945919896606. Epub 2019 Dec 22. PMID 31868125
- [Background] Klein CJ, Dalstrom MD, Weinzimmer LG, Cooling M, Pierce L, Lizer S. Strategies of Advanced Practice Providers to Reduce Stress at Work. Workplace Health Saf. 2020 Sep;68(9):432-442. doi: 10.1177/2165079920924060. Epub 2020 Jun 3. PMID 32491978
- [Background] Klein CJ, Weinzimmer LG, Dalstrom M, Lizer S, Cooling M, Pierce L. Investigating practice-level and individual factors of advanced practice registered nurses and physician assistants and their relationship to resilience. J Am Assoc Nurse Pract. 2021 Jul 29;34(2):310-321. doi: 10.1097/JXX.0000000000000639. PMID 34334766
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Result] Dyrbye LN, Johnson PO, Johnson LM, Halasy MP, Gossard AA, Satele D, Shanafelt T. Efficacy of the Well-Being Index to identify distress and stratify well-being in nurse practitioners and physician assistants. J Am Assoc Nurse Pract. 2019 Jul;31(7):403-412. doi: 10.1097/JXX.0000000000000179. PMID 30829967
- [Result] Klein CJ, Riggenbach-Hays JJ, Sollenberger LM, Harney DM, McGarvey JS. Quality of Life and Compassion Satisfaction in Clinicians: A Pilot Intervention Study for Reducing Compassion Fatigue. Am J Hosp Palliat Care. 2018 Jun;35(6):882-888. doi: 10.1177/1049909117740848. Epub 2017 Nov 23. PMID 29169248